CLINICAL TRIAL: NCT01677793
Title: Developmental Trajectory of Brain Structural Connectivity and Cognitive Function From Childhood to Adulthood
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Health Research Institutes, Taiwan (Other)
Responsible Party: Principal Investigator, Statistical Center, NTUHCTC, Susan Shur-Fen Gau, National Taiwan University Hospital
Other Study IDs: 201105115RC
Record Dates: First submitted 2012-08-30; First posted 2012-09-03 (Estimated); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Brain Structural Connectivity; Cognitive Function

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Child and adolescent population

SUMMARY:
Magnetic resonance imaging (MRI) is a premier modality to investigate structures and functions of human brain. In studies of children and adolescents, noninvasiveness of MRI makes it especially applicable. Developmental trajectory of gray matter volume and cortical thickness has been well studied in western countries. However, significant variability of brain structure has been reported between Chinese and Caucasian, and the variation may also exist in developmental trajectory of the brain. However, the maturation processes of neural fiber tracts in white matter are less understood. Diffusion tensor imaging (DTI), which has been frequently used to investigate the integrity of fibertracts in the literature, is limited in dealing with crossing fibers. Diffusion spectrum imaging (DSI) is a newly developed technique to improve the resolution of crossing fibers, and it is more suitable for detailed tractography assessment. In addition to establishing the template of brain structure (T1 and T2) and structural connectivity of our child, adolescent, and young adult population, the study has the following three aims.

1. To describe gender effect and developmental change of brain volume of different cortical and subcortical regions, thickness of cortex brain, and structural connectivity (e.g., frono-striatal, fronto-pareital, fronto-temporal and fronto-cerebeller tracts and superior longitudinal fasciculus II) across childhood through adolescent to adulthood;
2. To examine the gender effects and developmental change of attention, executive function and visual memory from childhood to adulthood and whether gender moderates these developmental changes; and
3. To correlate the structural connectivity and brain size and neuropsychological function within the same subjects.

DETAILED DESCRIPTION:
The investigators plan to recruit 140 healthy volunteers (70 males and 70 females), ages 8-21 without current and past history of any psychiatric disorder and autistic symptoms. All the participants will receive psychiatric interviews (K-SADS-E/SADS) and complete the Chinese AQ or SRS to screen for any psychiatric disorder or autistic symptoms. They will receive the WAIS-III or WISC-III (depending on their age) first to ensure their full-scale IQ greater than 80, followed by the CPT and CANTAB for a wide range assessments of attention, executive functions, and memory. The MRI assessments (T1 and T2 imaging, DSI, and resting-state fMRI) will be subsequently arranged within 2 weeks after psychiatric/neuropsychological assessments.

The investigators anticipate that this study (1) will establish the first template of brain anatomy and structural connectivity of children and adolescents in our population, (2) will be the first report on the developmental trajectory of brain of Chinese in both brain gross anatomy and tractography; (3) will provide evidence about how these development in brain structures associated with maturation in cognitive functions.

ELIGIBILITY:
Inclusion Criteria:

* Ages 8-21 without current and past history of any psychiatric disorder and autistic symptoms.

Exclusion Criteria:

* Current symptoms or lifetime history of DSM-IV-TR diagnosis of attention-deficit/hyperactivity disorder, pervasive developmental disorder, schizophrenia, schizoaffective disorder, delusional disorder, other psychotic disorder, organic psychosis, bipolar disorder, depression, severe anxiety disorders or substance use.
* With neurodegenerative disorder, epilepsy, involuntary movement disorder, congenital metabolic disorder, brain tumor, history of severe head trauma, and history of craniotomy.
* With major systemic disease.
* Full-scale IQ < 80.

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The sample consists of 140 healthy volunteers (70 males and 70 females). The ranges of age are 8-21 (around 5 males and 5 females in each age group). They will be recruited from schools and colleges.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Shur-Fen Gau, MD, PhD, Principal Investigator — National Taiwan University Hospital & College of Medicine
Locations (1):
- National Taiwan Univeristy Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Chiang HL, Chen YJ, Shang CY, Tseng WY, Gau SS. Different neural substrates for executive functions in youths with ADHD: a diffusion spectrum imaging tractography study. Psychol Med. 2016 Apr;46(6):1225-38. doi: 10.1017/S0033291715002767. Epub 2016 Jan 8. PMID 26744120
- [Derived] Chiang HL, Chen YJ, Lo YC, Tseng WY, Gau SS. Altered white matter tract property related to impaired focused attention, sustained attention, cognitive impulsivity and vigilance in attention-deficit/ hyperactivity disorder. J Psychiatry Neurosci. 2015 Sep;40(5):325-35. doi: 10.1503/jpn.140106. PMID 25871496